CLINICAL TRIAL: NCT02569034
Title: Dissociating Components of Anhedonia: Pilot Behavioral and fMRI Data for the Effort Expenditure for Rewards Task
Brief Title: Dissociating Components of Anhedonia: A Pilot fMRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB201400639-N; 5R03MH109336-02 (NIH); R03MH109336-01A1 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young Adults (Active Comparator): These participants will perform the Effort-Expenditure for Rewards Task (EEfRT) while an functional magnetic resonance imaging (fMRI) is performed. They will also complete a battery of both cognitive and anhedonia questionnaires.
  Interventions: Other: Functional Magnetic Resonance Imaging; Other: Effort-Expenditure for Rewards Task
- Older Adults (Experimental): These participants will perform the Effort-Expenditure for Rewards Task (EEfRT) while an functional magnetic resonance imaging (fMRI) is performed. They will also complete a battery of both cognitive and anhedonia questionnaires.
  Interventions: Other: Functional Magnetic Resonance Imaging; Other: Effort-Expenditure for Rewards Task

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging — Both groups will have the fMRI performed once. The fMRI will be use to to dissociate activity associated with both reward "wanting" and reward "liking" using the EEfRT. Learning more about the brain basis of components of anhedonia in both young and older adults is important in the context of previous research showing that risk-taking behavior and reward sensitivity changes with age, enhancing the knowledge of anhedonia.
  Other Names: fMRI
Other: Effort-Expenditure for Rewards Task — Both groups with have the EEfRT performed once. The EEfRT is an effort-based decision-making task that measures reward "wanting", in contrast to commonly used anhedonia questionnaires, which focus on reward "liking." This novel task may provide a useful measure of components of anhedonia in older adults and in different patient populations.
  Other Names: EEfRT

SUMMARY:
Anhedonia, decreased motivation for and sensitivity to rewarding experiences, is present in at least 1/3 of community dwelling older adults and is a feature of various psychiatric and neurological disorders, including late-life depression and Parkinson's disease. Anhedonia is associated with cognitive deficits, as well as poor clinical outcomes and increased mortality. Recent research suggests that anhedonia comprises motivational (reward "wanting") and consummatory (reward "liking") aspects. However, previous research on anhedonia has failed to dissociate these components, which may explain the contradictory findings in the literature. Recently, the Effort-Expenditure for Rewards Task (EEfRT) was developed in an effort to dissociate reward components in anhedonia. The EEfRT is an effort-based decision-making task that measures reward "wanting", in contrast to commonly used anhedonia questionnaires, which focus on reward "liking." This novel task may provide a useful measure of components of anhedonia in older adults and in different patient populations. Thus far no data is available on this task in elderly individuals, and the cognitive and neural correlates of components of the task have not been investigated. Given the paucity of research on the neurobiology of anhedonia, cognitive neuroscience studies using this task could fill a gap in the literature. The investigators are developing a line of cognitive neuroscience studies examining anhedonia in community-dwelling older adults and in late-life depression and Parkinson's disease. This study will involve gathering pilot behavioral and functional magnetic resonance imaging (fMRI) data in young and older adults performing the EEfRT task. Understanding the brain mechanisms underlying anhedonia in older adults and in different patient populations will have a translational impact by elucidating biological targets for treatment.

DETAILED DESCRIPTION:
Twenty young adults (aged 18-38) and 20 older adults (aged 60-80) will perform the EEfRT while fMRI data are acquired. To quantify brain activity associated with reward "wanting," the fMRI activation will be measured while participants view information about reward probability and choose to perform the easy or hard task, with greater reward associated with the hard task. The investigators will measure activation during presentation of reward magnitude to capture brain activity associated with reward "liking." Participants will also complete a brief cognitive battery and anhedonia questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-38 or 60-80 years
* Able to provide verbal and written consent
* Right-handed
* Native English speaker
* At least 12 years of formal education

Exclusion Criteria:

* Significant cognitive disturbance
* Self-report of current or past history of psychiatric disturbance other than major depression (e.g., bipolar disorder, schizophrenia, alcohol and/or substance abuse)
* Self-report of neurological disturbance (stroke, dementia, traumatic brain injury), chronic medical illness (HIV, metastatic cancer), or unstable medical conditions (cardiac or pulmonary disease)
* Physical impairments, language comprehension deficits, or significant hearing disturbances that would limit ability to perform tasks
* Current anticholinergic, psychotropic (stimulants or dopamine agonists), or anti-epileptic use
* Visual acuity difficulties that would interfere with task performance
* Motor deficits that may interfere with the use of the dominant hand for performance of button press associated with the EEfRT task
* MRI contraindications (e.g., ferrous metal in the body, claustrophobia, pregnancy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
fMRI Activity | Approximately Day 14 (Visit 2)
  To quantify brain activity associated with reward "wanting," the investigators will contrast fMRI activation while participants view information about reward probability and choose to perform the easy or hard task with activity during fixation. The investigators will contrast activation during performance feedback and presentation of reward magnitude with activation during fixation to capture brain activity associated with reward "liking." Parameter estimates (ß) will be generated, which indicated relative strength of covariance between the data and the hemodynamic response function (HRF). The investigators will use a three-dimensional spatial contiguity threshold of 20 voxels and a statistical significance threshold of p ≤ .005 to decrease the likelihood of spurious findings.
EEfRT Task Test | Approximately Day 14 (Visit 2)
  The EEfRT is a computerized task in which participants are presented with a series of repeated trials during which they choose between performing a ''hard-task'' or an ''easy-task'' in order to earn varying amounts of monetary rewards.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline (Visit 1)
  Cognitive screening instrument. The highest possible score is 30. 18 - 26 = mild cognitive impairment, 10 - 17 = moderate cognitive impairment and less than 10 = severe cognitive impairment.
Dementia Rating Scale-2 (DRS-2) | Baseline (Visit 1)
  The scale includes 36 tasks which are grouped into five subscales assessing different cognitive domains, namely: Attention, Initiation/Perseveration (I/P), Construction, Conceptualization and Memory.
Card Stroop Task | Baseline (Visit 1)
  Participants must 1) read color words (red, green and blue) aloud, 2) name the ink color of a string of X's presented in rows on a page, and 3) name the ink color of color words (red, green, blue) written in either the same or a different color as the word meaning.
Letter-Number Sequencing (Wechsler Adult Intelligence Scale, 4th Edition) | Baseline (Visit 1)
  Subjects hear a string a numbers and letters and must repeat them with the numbers first, in order, followed by the letters in alphabetical order.
Trail Making Test Parts A and B | Baseline (Visit 1)
  The task requires a subject to 'connect-the-dots' of 25 consecutive targets on a sheet of paper or computer screen. There are two parts to the test: A, in which the targets are all numbers (1,2,3..) and the test taker needs to connect them in sequential order, and B, in which the subject alternates between numbers and letters (1, A, 2, B, etc.). The test should be finished as quickly as possible within 5 minutes. The poorer the performance the higher the impairment.
Wisconsin Card Sorting Test | Baseline (Visit 1)
  A number of stimulus cards are to be match within 20 minutes. Participants must figure out the sorting rule based on feedback from the examiner.
Controlled Oral Word Association/Category Fluency | Baseline (Visit 1)
  Subjects are asked to name as many words as they can in 60 seconds based on either a letter (F, A, and S) or a category (animals) rule.
Digit Span (Wechsler Adult Intelligence Scale, 4th Edition) | Baseline (Visit 1)
  Subjects repeat a string of numbers in either the same order (digits forward) or in reverse order (digits backward).
California Verbal Learning Test II (CVLT-II) | Baseline (Visit 1)
  Subjects are asked to learn and remember a 16-item word list.
Brief Visuospatial Memory Test-Revised (BVMT-R) | Baseline (Visit 1)
  Subjects are asked to learn and remember the identity and location of 6 simple figures displayed on a page.
Temporal Experience of Pleasure scale (TEPS) | Baseline (Visit 1)
  18-item self-report questionnaire assessing anticipatory pleasure and consummatory pleasure
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline (Visit 1)
  The SHAPS measures hedonic capacity. A higher total SHAPS score will indicate a higher level of anhedonia or the inability to experience pleasure.
Positive Affect Negative Affect Scale (PANAS) | Baseline (Visit 1)
  Subjects are required to respond to a 20-item test using 5-point scale that ranges from very slightly or not at all (1) to extremely (5).
Beck Depression Inventory, 2nd Edition (BDI-II) | Baseline (Visit 1)
  21-item self-report questionnaire assessing symptoms of depression.
Geriatric Depression Scale (GDS) | Baseline (Visit 1)
  Subjects answer 30 yes/no questions assessing symptoms of depression.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline (Visit 1)
  This is a 20-item measure of depression severity.
State-Trait Anxiety Inventory (STAI) | Baseline (Visit 1)
  The STAI measures two extremes of anxiety affect, labeled state anxiety (A-State), and trait anxiety (A-Trait). Higher scores suggest higher levels of anxiety.
Apathy Scale (AS) | Baseline (Visit 1)
  14-item self-report questionnaire assessing symptoms of apathy over the previous 2-4 weeks
Lille Apathy Rating Scale (LARS) | Baseline (Visit 1)
  33 queries belonging to nine domains, each corresponding to a clinical manifestation of apathy

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Woods, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States